CLINICAL TRIAL: NCT01780584
Title: Oral Triiodothyronine Normalizes T3 Levels After Surgery For Pediatric Congenital Heart Disease
Brief Title: Can Oral T3 Normalize Thyroid Hormone Levels Following Cardiopulmonary Bypass in Children?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Eva M Marwali,MD, Pediatric Cardiac Intensivist, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LB05.01/1.4/235/2010
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Low T3 Syndrome
Keywords: congenital heart surgery, thyroid hormones
MeSH Terms: conditions — Euthyroid Sick Syndromes | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral T3 low dose & placebo (Active Comparator): Oral T3 low dose administer through nasogastric tube 0.5 mcg/kg (max 10 mcg) starting on induction of anesthesia and then every 24 hours alternating with placebo, which was given 12 hours after the first dose of oral T3 and then every 24 hours until 60 hours post anesthesia induction (3 doses oral T3, 3 doses placebo)
  Interventions: Drug: Oral T3 Low dose; Drug: Placebo
- Placebo (Placebo Comparator): Placebo (saccharin lactic) administer through nasogastric tube, given starting on induction of anesthesia and then every 12 hours until 60 hours post-anesthesia induction (6 doses total)
  Interventions: Drug: Placebo
- Oral T3 high dose (Experimental): Oral T3 high dose administer through nasogastric tube 0.5 mcg/kg (max 10 mcg) q12h starting on induction of anesthesia until 60 hours post-anesthesia (6 doses oral T3)
  Interventions: Drug: Oral T3 high dose

INTERVENTIONS:
Drug: Oral T3 Low dose — Comparison of different dosages of drug. Low dose group oral T3 is 0.5 mcg/kg q24h
  Other Names: Tetronine
  Arms: Oral T3 low dose & placebo
Drug: Placebo — Comparison of different dosages of drug. In low dose group, placebo was given alternately with oral T3 every 12h with a total 3 doses for placebo and 3 doses for oral T3
  Other Names: Sacharin Lactis
  Arms: Oral T3 low dose & placebo; Placebo
Drug: Oral T3 high dose — Comparison of different dosages of drugs. Oral T3 high dose is 0.5 mcg/kg q12h
  Other Names: Tetronine
  Arms: Oral T3 high dose

SUMMARY:
Low triiodothyronine (T3) syndrome defines as decrease of T3 levels during critically ill. This decrease of T3 levels was observed after congenital heart surgery using cardiopulmonary bypass. Previous largest study,Triiodothyronine for Infants and Children Undergoing Cardiopulmonary bypass (TRICC) study showed T3 supplementation decreased time to extubation for infants less than 5 months undergoing cardiopulmonary bypass. Intravenous regiment was known effective in maintaining T3 levels during pediatric cardiac surgery. This drug preparation however is not commonly used in many countries due to the relatively high costs and/or the simple lack of availability. The use of oral T3 to treat postoperative low T3 levels in pediatric patients has not been reported so far, although recent adult studies showed benefit in using oral T3 after cardiac surgery. The purpose of this study was to determine if oral T3 supplementation could prevent the decline of serum T3 in children less than 2 years of age undergoing congenital heart surgery using CPB.

DETAILED DESCRIPTION:
The Research Ethics Board at the National Cardiovascular Center Harapan Kita approved this study and written, informed consent was obtained from the parents or legal guardians before randomization. Randomization by block permutation was performed to determine treatment group assignment. Randomization occured on the day before surgery by a nurse investigator. A pharmacist who was not involved in the study prepared the study medication. Investigators and participants were blinded to the assigned group until after the end of the study.

Thyroid hormonal levels were analyzed by standard 3rd generation thyrotropic-stimulating hormone (TSH), serum free T4 (FT4), free T3 (FT3), and total T3 (TT3) Micro particle Enzyme Immunoassays (Abbott Laboratories, Abbott Park, USA). The serum total T4 (TT4) assay used a Fluorescence Polarization Immunoassay (Abbott Laboratories, Abbott Park, USA). Hormone levels were measured on induction of anesthesia, before the study drug was given (T0) and at 1, 6, 18, 36 and 72 hours after removal of the aortic-cross-clamp.

Baseline clinical data collected included age, gender, birth weight, type of operation, and Aristotle score. Diagnosis and operative procedures were classified as high or low risk with an Aristotle score cut off of ≥ 9 as high risk. As modifying factors, we measured duration of surgery, cardiopulmonary bypass (CPB) time, cross-clamp time, ultrafiltration during CPB and degree of hypothermia during CPB, and the use of amiodarone. Non-pulsatile perfusion technique was used during CPB. Steroid (methyl prednisolone 35-50 mg/kg) was given before CPB. We used povidone-iodine for skin disinfection in all subjects. Although this study was not powered to detect clinical differences between the treatment groups, clinical outcome parameters were measured as a potential guide to subsequent adequately powered larger treatment studies. Serum lactate was measured at 1 hour, 4 hours and day 1 post surgery. Hemodynamic monitoring included heart rate, heart rhythm, and blood pressure which were recorded hourly for the first 6 hours then every 6 hours until 72 hours after surgery. Overt symptoms of hyperthyroidism were grounds for immediate removal of the subjects from the study. Time to extubation and length of stay in the intensive care unit and hospital were recorded.

Statistical analysis and sample size: The primary efficacy analysis assessed the difference between the treatment (high-dose, low-dose) and control groups with regard to the effect of T3 supplementation on the measured TT3 and FT3 serum levels. We anticipated a difference of 2.0 pg/ml in FT3 with a standard deviation of 0.8 pg/ml between groups. For a statistical power of 80% to identify a treatment effect and at a level of significance of 0.05 ( 2-sided), the target total sample size was 45 subjects, with 15 in each treatment group. Demographic data, safety and clinical outcomes were compared using the X2 test. Continuous variables for characteristics and outcomes were analyzed using one way ANOVA for data with normal distribution or the Kruskal Wallis test for not normally distributed data. Repeated measures ANOVA was used to analyze all thyroid hormone levels and clinical outcomes for those variables that were measured repeatedly over time. Paired Student's t-test for parametric or Wilcoxon signed rank test for non-parametric tests were used to evaluate the mean difference of hormone levels and clinical outcomes over time in each treatment group. Statistical significance was defined by p-values less than 0.05. Descriptive statistics are reported as mean ± standard error of the mean.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 0-2 years of age
* Aristotle score of 6 and above
* underwent cardiac surgery using cardiopulmonary bypass

Exclusion Criteria:

* birth weight less than 2 kg for neonates
* preoperative tachyarrhythmia or need for anti arrhythmic treatment
* clinical sepsis confirmed by culture
* preoperative renal insufficiency
* known thyroid and metabolic disorder
* any contraindication for oral T3 administration

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Marwali, MD, Principal Investigator — Pediatric Cardiac ICU National Cardiovascular Center Harapan Kita Jakarta
Locations (1):
- Pediatric Cardiac ICU National Cardiovascular Center Harapan Kita Jakarta, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Result] Portman MA, Slee A, Olson AK, Cohen G, Karl T, Tong E, Hastings L, Patel H, Reinhartz O, Mott AR, Mainwaring R, Linam J, Danzi S; TRICC Investigators. Triiodothyronine Supplementation in Infants and Children Undergoing Cardiopulmonary Bypass (TRICC): a multicenter placebo-controlled randomized trial: age analysis. Circulation. 2010 Sep 14;122(11 Suppl):S224-33. doi: 10.1161/CIRCULATIONAHA.109.926394. PMID 20837917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruitment was done from Pediatric Cardiac Intensive Care Unit at the National Cardiovascular Center Harapan Kita, Jakarta, Indonesia between April, 2010 and September, 2010.
Pre-assignment Details: There were 47 individuals screened for participation, and consent to participate was obtained from 46 (98%). One subjects from whom did not participate because of surgical postponement. A total of 45 subjects were randomized to 3 groups of 15.
Groups:
- Oral T3 Low Dose: Oral T3 low dose administer through nasogastric tube 0.5 mcg/kg (max 10 mcg) starting on induction of anesthesia and then every 24 hours alternating with placebo, which was given 12 hours after the first dose of oral T3 and then every 24 hours until 60 hours post anesthesia induction (3 doses oral T3, 3 doses placebo)
Period: Overall Study
Arm/Group | Placebo | Oral T3 Low Dose | Oral T3 High Dose
Started | 15 | 15 | 15
Completed | 14 | 14 | 13
Not Completed | 1 | 1 | 2
Not completed — Death | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject in in oral T3 low dose group with hypertension due to unrecognized coarctation and one subject in oral T3 high dose group with inability to attain enteral feeds were withdrawn from the treatment protocol. Therefore there were 43 subjects included in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral T3 Low Dose | Placebo | Oral T3 High Dose | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 15 | 45
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.9 (0.5) | 0.8 (0.4) | 0.8 (0.6) | 0.9 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 9 | 25
  Male | 9 | 5 | 6 | 20
Region of Enrollment [Number; unit: participants]
  Indonesia | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Free T3 (FT3) Levels
Description: Free T3 levels were measured up to 36 hours after cross-clamp removal
Time Frame: during the first 36 hours after cross clamp removal
Population: Two subjects (one in T3 low dose and one in T3 high dose) were withdrawn from the treatment protocol. The withdrawal in low dose group was because of severe hypertension caused by a previously unrecognized coarctation of the aorta, and the high dose group withdrawal was due to massive gastrointestinal bleeding.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo | Oral T3 Low Dose | Oral T3 High Dose
Number analyzed (Participants) | 15 | 14 | 14
pg/ml
  hour 0 | 3.6 (0.4) | 4.5 (0.6) | 3.9 (0.2)
  hour 1 | 3.6 (0.3) | 4.1 (0.5) | 4.3 (0.2)
  hour 6 | 2.9 (0.3) | 3.3 (0.3) | 3.7 (0.3)
  hour 18 | 2.4 (0.2) | 2.6 (0.4) | 3.8 (0.4)
  hour 36 | 1.6 (0.2) | 2.1 (0.3) | 4.4 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Oral T3 Low Dose vs Oral T3 High Dose; Null hypothesis: no difference of free T3 (FT3) levels will be found between placebo, low dose and high dose group. We anticipated a difference of 2 pg/ml in FT3 with a standard deviation of 0.8 pg/ml between groups. For a statistical power of 80% to identify a treatment effect and at a level significance of 0.05 (2-sided); Test type: Superiority or Other; p < 0.05, ANOVA — Repeated Anova was used to determine whether there was difference of FT3 levels between groups; Mean Difference (Final Values) = 2, 95% CI 2-sided [1 to 3], Standard Error of Mean 0.8

2. Secondary Outcome: Number of Patients With Possible Side Effects of Thyroid Hormone Supplementation Particularly Suggesting Hyperthyroid Symptoms.
Description: Specific symptoms of hyperthyroidism included cardiac dysrhythmia requiring medical or electrical treatment, hypertension (mean systolic or diastolic blood pressure more than 2 standard deviation above normal for age) and hyperthermia (>37.5 degree Celsius). One patient in low dose group had hypertension directly after surgery due to unrecognized coarctation of the aorta and this patient was withdrawal from the protocol.
Time Frame: Since the first dose of oral T3 until 7 days after surgery
Population: Three patients were excluded from adverse effect analysis. Two patients, each in placebo and high dose group were on Extracorporeal Membrane Oxygenation. One patient in high dose group could not attained enteral feeds due to gastrointestinal bleeding and was withdrawal from the protocol.
Measure: Number; unit: participants
Arm/Group | Placebo | Oral T3 Low Dose | Oral T3 High Dose
Number analyzed (Participants) | 14 | 15 | 13
participants | 0 | 1 | 0

3. Other Pre Specified Outcome: Postoperative Time to Extubation
Description: Postoperative time to extubation is length of time on ventilator.
Time Frame: up to 3 months after surgery
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Oral T3 Low Dose | Oral T3 High Dose
Number analyzed (Participants) | 14 | 14 | 13
hours | 23 [15 to 144] | 36.5 [5 to 794] | 17 [8 to 224]
Statistical Analysis 1: Comparison: Placebo vs Oral T3 Low Dose vs Oral T3 High Dose; Null hypothesis: no difference of time to extubation between group. Statistical power 80% and level of significance 0.05; Test type: Superiority or Other; p = 0.31, Kruskal-Wallis — Kruskal Wallis test was used to determine any difference of time of extubation between groups; Median Difference (Final Values) = 5, 95% CI [3 to 10]

4. Other Pre Specified Outcome: Postoperative Length of Stay in Intensive Care Unit
Time Frame: up to 3 months after surgery
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | Oral T3 Low Dose | Oral T3 High Dose
Number analyzed (Participants) | 14 | 14 | 13
hours | 48.5 [20 to 258] | 109.5 [22 to 816] | 87 [22 to 456]
Statistical Analysis 1: Comparison: Placebo vs Oral T3 Low Dose vs Oral T3 High Dose; Null hypothesis: there is no difference of length of stay in Intensive Care Unit. Statistical power 80% and level of significance 0.05; Test type: Superiority or Other; p = 0.4, Kruskal-Wallis; Median Difference (Net) = 50, 95% CI [40 to 60]

5. Other Pre Specified Outcome: Postoperative Hospital Length of Stay
Time Frame: up to 3 month after surgery
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | Oral T3 Low Dose | Oral T3 High Dose
Number analyzed (Participants) | 14 | 14 | 13
days | 6 [5 to 26] | 17.5 [2 to 34] | 10 [5 to 41]
Statistical Analysis 1: Comparison: Placebo vs Oral T3 Low Dose vs Oral T3 High Dose; Null hypothesis: there is no difference of postoperative hospital length of stay between groups. Statistical power 80% and level of significance 0.05; Test type: Superiority or Other; p = 0.06, Kruskal-Wallis; Median Difference (Final Values) = 10, 95% CI [5 to 15]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Serious adverse events was defined as mortality within 3 months. Other adverse events were symptoms of suspected of hyperthyroidism that observed within 7 days since the study started.
Arm/Group | Oral T3 Low Dose | Placebo | Oral T3 High Dose
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 1/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral T3 Low Dose (N=15) | Placebo (N=15) | Oral T3 High Dose (N=15)
Mortality (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) — One patient in placebo group and one patient in high dose group were died during 7 days after surgery, due to irreversible cardiac pump failure. One patient in low dose group was died due to sepsis and heart failure 34 days after surgery.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral T3 Low Dose (N=15) | Placebo (N=15) | Oral T3 High Dose (N=15)
Symptoms of suspected hyperthyroidism (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Symptoms suggested hyperthyroidism were observed within 7 days after surgery. One patient in low dose group had hypertension after surgery due to unrecognized coarctation of the aorta.

LIMITATIONS AND CAVEATS:
The lack of power to detect differences in clinical outcomes. There was also insufficient power to detect potentially subtle adverse effects of T3 supplementation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No